CLINICAL TRIAL: NCT03832218
Title: Executive Function Disorders and Anxio-depressive Symptomatology in Children and Adolescents With Mitochondrial Pathologies
Acronym: MITOPSY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 49RC19_0004
Record Dates: First submitted 2019-02-01; First posted 2019-02-06 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-04

CONDITIONS: Mitochondrial Diseases
MeSH Terms: conditions — Mitochondrial Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mitochondrial disease (Other): Psychiatric assessment
  Interventions: Diagnostic Test: Psychiatric assessment

INTERVENTIONS:
Diagnostic Test: Psychiatric assessment — Psychiatric assessment and neuropsychological tests
  * Test : Wechsler Intelligence Scale for Children (WISC-V)
  * Test :Behavior Rating Inventory of Executive Function (BRIEF) : BRIEF-Parents, BRIEF-Teacher
  * Global Assessment of Functioning Scale
  * Scale : Brief Psychiatric Rating Scale (BPRS)
  * Test : Children Depression Inventory (CDI)
  * Scale : Revised-Children's Manifest Anxiety Scale (R-CMAS)
  * Survey : Pediatric Quality of Life Inventory Version 4.0 (PedsQL™ 4.0)
  * Scale : Conners' scale (parents and teachers)

SUMMARY:
The major steps forward of the neurosciences in recent years have linked psychiatric diseases, neuropsychological symptoms and brain dysfunctions. The cerebral functioning requiring a big quantity of energy, mitochondria, essential organelles in the cellular energy processes, are at present considered as a way of research for big interest in neurology and in psychiatry. Thus, an increasing number of studies describe potential links between mitochondrial dysfunction and psychiatric symptomatology. The clinical symptomatology of children with mitochondrial cytopathy is varied. Well described neurologically and somatically, it is significantly less in its psychiatric aspects. However, psychiatric symptoms are frequently associated and this symptom has already been described in adult patients. The symptoms mainly include depressive and anxiety disorders, or even tables suggestive of psychotic disorders, which would precede the diagnosis of mitochondrial disease of 13 years on average.

Neuropsychological disorders refer to disorders of the higher functions following a cerebral anomaly (language, praxis, motricity, gnosis, visual spatial processing, memory, attention, intelligence, executive functions ...). Tests validated in French and adapted to children and adolescents can identify neuropsychological disorders in these populations.

ELIGIBILITY:
Inclusion Criteria:

* Child with mitochondrial cytopathy (defined by the presence of a mutation known to cause mitochondrial cytopathy or mitochondrial respiratory chain abnormality)
* Aged 6 to 17 years
* Beneficiary of a Social Security regime
* Parents sign consent

Exclusion Criteria:

* Child refusal to participate in the study
* Complete inability to complete questionnaires (e.g. non-communicating child)
* Child already included in intervention research modifying care

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2019-05-02 (Actual); Primary Completion 2020-02-27 (Actual); Study Completion 2020-02-27 (Actual)

PRIMARY OUTCOMES:
Prevalence of the psychiatric disorders in a population of children reached of mitochondrial disease | Day 1
  Psychiatric assessment and neuropsychological tests
  Test : Wechsler Intelligence Scale for Children (WISC-V) Test :Behavior Rating Inventory of Executive Function (BRIEF) : BRIEF-Parents, BRIEF-Teacher Global Assessment of Functioning Scale Scale : Brief Psychiatric Rating Scale (BPRS) Test : Children Depression Inventory (CDI) Scale : Revised-Children's Manifest Anxiety Scale (R-CMAS) Survey : Pediatric Quality of Life Inventory Version 4.0 (PedsQL™ 4.0) Scale : Conners' scale (parents and teachers)

CONTACTS AND LOCATIONS:
Locations (1):
- Dr RIQUIN Elise, Angers, France

IPD SHARING:
Plan to Share IPD: Undecided